CLINICAL TRIAL: NCT06564285
Title: The Effects of a Novel Nutritional Product on Nutrient Gaps and Gut Health in Adults With Occasional Gastrointestinal Issues
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Athletic Greens International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: AG-AG1-53-09
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Gastrointestinal Microbiome; Nutrition, Healthy

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Placebo Controlled Design
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Maltodextrin + Flavoring
  Interventions: Dietary Supplement: Placebo
- AG1 - Nutritional Supplement (Experimental): A foundational nutritional supplement consisting of vitamins, minerals, probiotics, prebiotics, and whole food ingredients
  Interventions: Dietary Supplement: AG1 - Nutritional Supplement

INTERVENTIONS:
Dietary Supplement: AG1 - Nutritional Supplement — A foundational nutritional supplement consisting of vitamins, minerals, probiotics, prebiotics, and whole food ingredients
  Arms: AG1 - Nutritional Supplement
Dietary Supplement: Placebo — Maltodextrin placebo
  Arms: Placebo

SUMMARY:
This study is a randomized, double-blind, placebo-controlled study of N=40 adult men and women with occasional GI issues. This study to assess the effect of a novel dietary supplement on the gut microbiome, nutrient gaps, and tolerability.

ELIGIBILITY:
To be eligible to participate in this study, an individual must meet all of the following criteria:

* Provide voluntary signed and dated informed consent.
* Does not have any chronic health conditions that could impact participation in this study such as oncological or psychiatric disorders.
* No known history of chronic illness or disease.
* Aged between 18 and 60 years (inclusive).
* Body Mass Index of 20-34.9 (inclusive).
* Agree to maintain existing dietary and physical activity patterns throughout the study period.
* Willing and able to comply with the study protocol.
* Self-reported gastrointestinal symptoms, such as self-reported abdominal pain, gas and bloating after meals, heartburn/acid reflux after meals, and issues with digestion.
* Must be in good general health.
* Following a stable, consistent diet pattern.
* Agree to refrain from any lifestyle changes that may affect their GI tract and IBS symptoms for the duration of the study.
* Not currently taking and not planning on introducing any product, supplement or medication aimed at gut health or nutritional gaps during the study period.
* Resides in the United States.

An individual who meets the following criteria will be excluded from participation in this study:

* Prior prescriptions for IBS or any other medication (OTC and prescription) targeting the gut.
* Taking any supplements targeting the gut in the past 30 days.
* Current IBS treatment (e.g. proton pump inhibitors, laxatives).
* Follow an extreme diet intervention. This includes specific exclusion-type diets like vegan, vegetarian, carnivore, paleo, Atkins, ketogenic etc.
* Experienced significant weight loss (10% total body weight) in the past 3 months prior to study participation.
* Usage of any medication or herbal remedies which can affect the GI tract.
* Food intolerances/allergies.
* History of GI tract cancers.
* Celiac disease/gluten intolerance.
* Pregnant women, women trying to conceive, women less than 120 days postpartum, or nursing women.
* Anyone with any allergy requiring the use of an Epi-pen.
* Multivitamin/Multimineral supplement consumption within the past 3 months.
* History of use of medications or dietary supplements known to confound the study or its endpoints.
* History of unstable or new-onset cardiovascular, liver, or renal conditions.
* History of diabetes or endocrine disorder.
* Anyone who has received an antibiotic, antifungal, antiparasitic, or antiviral treatment within 90 days prior to the study.
* Excessive alcohol consumption (more than 2 standard alcoholic drinks per day or more than 10 drinks per week) within the past 6 months.
* Current smokers or smoking within the past month.
* History of drug abuse or dependence.
* History of hyperparathyroidism or an untreated thyroid condition.
* History of malignancy in the previous 5 years except for non-melanoma skin cancer (basal cell cancer or squamous cell cancer of the skin).
* Prior gastrointestinal bypass surgery (Lapband, etc.).
* Other known gastrointestinal or metabolic conditions that might impact nutrient absorption or metabolism, e.g., short bowel syndrome, IBS/IBD, diarrheal illnesses, history of colon resection, gastroparesis, and Inborn errors of metabolism (such as PKU).
* Diagnosed chronic inflammatory condition (e.g., rheumatoid arthritis, Crohn's, ulcerative colitis, Lupus, HIV/AIDS, etc.).
* Previous medical diagnosis of asthma, gout, or fibromyalgia.
* A change in hormone therapy, including oral contraceptives, within 4 weeks prior to screening, or unwilling to maintain current hormone therapy/oral contraceptive use throughout the course of the study.
* Known allergy or sensitivity to any ingredient in the test formulations as listed in the product label or in the placebo ingredients.
* Currently participating in another research study with an investigational product or have been in another research study in the past 30 days or planning on taking part in another research study during this study's duration.
* Has undergone any surgery or invasive treatments in the previous six months or has any planned for during the study period.
* Anyone taking any supplements that have the same ingredients as those in the test product.
* Has taken a probiotic, prebiotic, or postbiotic in the past 30 days.
* Currently taking any opioid medications such as oxycodone (OxyContin®), hydrocodone (Vicodin®), codeine, morphine, or kratom.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-08-28 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Gut Microbiome | 14 days
  Examine changes in the gut microbiome via fecal metagenomics and metabolomics

SECONDARY OUTCOMES:
Nutrient Gaps | 14 days
  Assess nutrient gaps by dietary record assessment utilizing The Automated Self-Administered 24-hour (ASA24®) Dietary Assessment Tool

OTHER OUTCOMES:
Digestive Tolerability | 14 days
  A Digestive Quality of Life Questionnaire (DQLQ) will be utilized to assess the effect of the interventions on participant's digestive health. Scores range from 0 to 9 with a higher score indicating worse digestion associated with quality of life
GI Tolerability | 14 days
  The Gastrointestinal Symptom Rating Scale will be provided to assess the effect of the intervention on GI symptoms. Scores range from 1 to 7 with a higher score indicating a higher level of discomfort

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No